CLINICAL TRIAL: NCT04136145
Title: An Open-label, Randomized, Parallel Group, Single Dose Study to Investigate the PK and Safety of Belimumab 200 mg Intravenous and 200 mg Subcutaneous Via Auto-injector in Chinese Healthy Participants
Brief Title: Single Dose Study to Investigate the Pharmacokinetics (PK) and Safety of Belimumab 200 Milligrams (mg) Intravenous and 200 mg Subcutaneous Via Auto-injector in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209629
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: belimumab; Chinese; intravenous; subcutaneous; auto-injector
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:2 ratio to receive one treatment of either IV or SC administration of belimumab 200 mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belimumab SC (Experimental): Subjects will be administered a single dose of belimumab 200 mg via the SC route. The dose will be administered in the front of the thigh via auto-injector device.
  Interventions: Drug: Belimumab for SC
- Belimumab IV (Experimental): Subjects will be administered a single dose of belimumab 200 mg via the IV route administered over approximately 1 hour.
  Interventions: Drug: Belimumab for IV

INTERVENTIONS:
Drug: Belimumab for IV — Belimumab will be available as white to off-white lyophilized cake at a unit dose strength of 400 mg to be reconstituted and diluted in normal saline to obtain 200 mg per dose.
  Arms: Belimumab IV
Drug: Belimumab for SC — Belimumab will be available as clear to opalescent, colorless to pale yellow sterile solution at unit dose strength of 200 mg/milliliter (mg/mL) for SC injection in a single-use, prefilled syringe contained within an auto-injector device.
  Arms: Belimumab SC

SUMMARY:
This is an open-label, randomized, parallel group, single dose study in healthy Chinese subjects. The purpose of this study is to characterize the pharmacokinetic profile and safety profile of 200 mg single dose of belimumab, administered either intravenously or subcutaneously via auto-injector. Each subject will be randomized in a 1:2 ratio to receive a single dose of either intravenous (IV) or subcutaneous (SC) administration of belimumab 200 mg. The total study duration will be approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.
* Chinese healthy male or female between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Healthy as defined as being free from clinically significant illness or disease as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital sign, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied, may be included only if the investigator (in consultation with the GlaxoSmithKline (GSK) medical monitor if necessary) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Non-smoker or ex-smoker having ceased smoking for at least 6 months.
* Body weight >=45.0 kilograms (kg) for females, >=50.0 kg for males, and body mass index (BMI) within the range 19.0<= to <=26.0 kilograms per meter square (kg/m^2).
* Both male and female subjects are eligible to participate.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: i) Not a woman of childbearing potential (WOCBP) OR ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 16 weeks after the last dose of belimumab.

Exclusion Criteria:

* A positive test for syphilis, positive Hepatitis C antibody, human immune deficiency syndrome (HIV) antigen/antibody, at Screening. For Hepatitis B: subjects with a positive hepatitis B surface antigen (HbsAg) and/or a positive anti-hepatitis B core (HBc) result will be excluded.
* A positive result of pre-study drug screen (including at minimum: amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines).
* ALT or AST >1.2 times upper limit of normal (ULN).
* Bilirubin >1.2 times ULN (isolated bilirubin >1.2 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTc >450 milliseconds (msec) based on single ECG. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine read or manually over-read.
* Immunoglobulin (M, A, G) level is <Lower limit of normal (LLN) at Screening.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of major organ transplant: e.g., heart, lung, kidney, liver, or hematopoietic stem cell transplant.
* History of malignant neoplasm within the last 5 years, except for adequately treated basal or squamous cell cancers of the skin, or carcinoma in situ of the uterine cervix.
* Subjects with a sitting position systolic blood pressure <90 millimeters of mercury (mmHg) or >=140 mmHg and/or a sitting diastolic blood pressure <50 mmHg or >=90 mmHg and/or systolic blood pressure drop from supine to standing of >30 mmHg.
* Symptomatic herpes zoster within 3 months prior to Screening.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posteroanterior) and a positive (not indeterminate) QuantiFERON-TB Gold test.
* History of any infection requiring hospitalization or treatment with antivirals, antibiotics, anti-fungals, anti-parasitic agents or vaccination within 30 days prior to the administration of study medication.
* History of regular alcohol consumption exceeding, on an average, 14 drinks/week for men or 7 drinks/week for female (1 drink = 5 ounces [150 mL] of wine or 350 mL of beer or 1.5 ounces [45 mL] of 80 proof distilled spirits) within 6 months of Screening.
* The subject had participated in a clinical study or post-marketing study with an investigational or a non-investigational product during the previous 4 months or 5 half-lives (whichever is longer) preceding the administration of study medication of this study.
* Exposure to more than 4 new chemical entities within 12 months prior to the dosing day.
* The subject planned to concurrently participate in another clinical study or post marketing study.
* Use of any prescription or non-prescription medications including vitamins, herbal and dietary supplements within the 14 days or 5 half-lives (whichever is longer) prior to the administration of study medication.
* History of B cell targeted therapy (rituximab, other anti-cluster of differentiation (CD)20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], B lymphocyte stimulator (BlyS)-receptor fusion protein [BR3], Transmembrane activator and calcium-modulator and cytophilin ligand interactor (TACI)-fusion (Fc), LY2127399 [anti-B cell-activating factor receptor (BAFF)] or belimumab) at any time.
* Have received a live vaccine within 30 days of Day 1 or anticipate receipt of a live vaccine during the study or within 120 days after the last dose administration of study drug.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy (excluding pollen allergy) without current symptoms.
* History of anaphylactic reaction to any food, drug, or insect bite/sting.
* History of allergic reaction to parenteral administration of contrast agents, foreign proteins, or monoclonal antibodies.
* Donation of blood or blood products or significant blood loss in excess of 400 mL within 4 months or 200 mL within 2 months prior to administration
* Subject is mentally or legally incapacitated, or unwillingness or inability (including mentally or legally incapacity) to follow the procedures outlined in the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Meng X, Wang Q, Wu S, Pu D, Zhang A, Fang S, Zhou X, Lu H. Pharmacokinetics and Safety of Intravenous and Subcutaneous Auto-injector Single-dose Belimumab in Healthy Chinese Volunteers: A phase 1, Randomized, Open-label Study. Rheumatol Ther. 2021 Dec;8(4):1711-1724. doi: 10.1007/s40744-021-00366-0. Epub 2021 Sep 23. PMID 34554352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, parallel group, single dose study to evaluate safety and pharmacokinetics (PK) of belimumab, administered either intravenously (IV) or subcutaneously (SC) via an auto-injector in healthy Chinese participants.
Pre-assignment Details: A total of 171 participants were screened and 36 participants were enrolled and randomized in the study.
Groups:
- Belimumab 200 mg IV: Healthy Chinese participants were administered a single IV infusion of belimumab at a dose of 200 milligram (mg), infused over approximately 1 hour.
- Belimumab 200 mg SC: Healthy Chinese participants were administered a single SC dose of belimumab 200 mg in the front of the thigh via an auto-injector device.
Period: Overall Study
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Started | 12 | 24
Completed | 12 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC | Total
Number analyzed (Participants) | 12 | 24 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.9 (3.99) | 29.1 (6.44) | 28.7 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 20 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 12 | 24 | 36

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentration of Belimumab Following Intravenous Administration
Description: Blood samples were collected at indicated time points for measurement of serum concentrations of belimumab following intravenous administration. Pharmacokinetic Population comprised of all safety participants (all randomized participants who received at least one dose of study treatment) for whom at least one evaluable pharmacokinetic sample was obtained and analyzed.
Time Frame: Pre-dose (prior to start of belimumab IV infusion), 30 minutes (after the start of infusion), 0 hour (end of infusion); at 1, 6, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344 and 1680 hours after end of infusion
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Belimumab 200 mg IV
Number analyzed (Participants) | 12
Nanograms per milliliter
  Pre-dose (prior to start of belimumab IV infusion) | 0.0 (0.00)
  30 minutes (after the start of infusion) | 26567.4 (3602.68)
  0 hour (end of infusion) | 63403.2 (6104.64)
  1hour after end of infusion | 64474.6 (9167.16)
  6 hours after end of infusion | 57450.1 (7804.49)
  24 hours after end of infusion | 50284.8 (4898.92)
  48 hours after end of infusion | 40738.2 (6858.36)
  72 hours after end of infusion | 32845.9 (9835.93)
  96 hours after end of infusion | 30995.0 (6472.10)
  168 hours after end of infusion | 23850.3 (3898.42)
  336 hours after end of infusion | 15930.7 (3859.50)
  504 hours after end of infusion | 11291.5 (3860.41)
  672 hours after end of infusion | 10115.7 (2289.97)
  1008 hours after end of infusion | 5838.3 (1868.93)
  1344 hours after end of infusion | 3146.7 (1275.16)
  1680 hours after end of infusion | 1916.6 (936.49)

2. Primary Outcome: Serum Concentration of Belimumab Following Subcutaneous Administration
Description: Blood samples were collected at indicated time points for measurement of serum concentrations of belimumab following subcutaneous administration.
Time Frame: Pre-dose and at 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours, 240 hours, 336 hours, 504 hours, 672 hours, 1008 hours, 1344 hours and 1680 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Belimumab 200 mg SC
Number analyzed (Participants) | 24
Nanograms per milliliter
  Pre-dose | 0.0 (0.00)
  6 hours post-dose | 963.8 (875.47)
  24 hours post-dose | 6255.4 (4255.21)
  48 hours post-dose | 11838.9 (5838.53)
  72 hours post-dose | 14501.9 (6105.54)
  96 hours post-dose | 16682.3 (6038.30)
  120 hours post-dose | 16131.3 (6055.17)
  144 hours post-dose | 16752.1 (5184.15)
  168 hours post-dose | 16825.5 (5095.95)
  240 hours post-dose | 17262.9 (3702.00)
  336 hours post-dose | 14724.2 (3519.94)
  504 hours post-dose | 11235.9 (2928.08)
  672 hours post-dose | 7551.1 (2836.06)
  1008 hours post-dose | 4720.3 (1827.40)
  1344 hours post-dose | 2651.6 (1345.36)
  1680 hours post-dose | 1365.7 (931.47)

3. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs were measured in a semi-supine position after five minutes of rest and included tympanic temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate. The normal ranges were: temperature (35.0-38.0 degrees celsius), SBP (85-160 millimeters of mercury [mmHg]), DBP (45-100 mmHg), heart rate (60-90 beats per minute). Number of participants with abnormality in any vital signs are presented. Safety Population comprised of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were recorded with the participants in a semi-supine position, after 5 minutes of rest using an ECG machine. Abnormal findings were categorized as clinically significant and not clinically significant. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of participants with clinically significant and not clinically significant abnormal ECG findings have been presented.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants
  Abnormal-Not Clinically significant | 3 | 7
  Abnormal-Clinically significant | 0 | 2

5. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The normal ranges were: alanine aminotransferase(7-40 international units per liter[IU/L]), albumin(40-55 grams per liter[g/L]), alkaline phosphatase(35-100 IU/L), amylase(25-125 units per liter), aspartate aminotransferase(13-35 IU/L), bilirubin(Bil.)(3.4-20.5 micromoles per liter [µmol/L]), calcium(2.1-2.55 millimoles per liter[mmol/L]), chloride(99-110 mmol/L), cholesterol(Chol.)(0-5.17 mmol/L), creatine kinase(29-168 IU/L), creatinine(41-73 µmol/L), direct Bil.(0-8.6 µmol/L), gamma glutamyl transferase(7-45 IU/L), glucose(3.9-6.1 mmol/L), high density Chol.(1.04-1.55 mmol/L), low density Chol.(2.59-4.11 mmol/L), lactate dehydrogenase(120-250 IU/L), phosphate(0.74-1.52 mmol/L), potassium(3.5-5.3 mmol/L), protein(65-85 g/L), sodium(137-147 mmol/L), triglycerides(0-1.69 mmol/L), urate(150-350 µmol/L), urea(2.6-7.5 mmol/L). Number of participants with abnormal clinical chemistry parameters are presented.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants | 12 | 24

6. Secondary Outcome: Number of Participants With Abnormal Hematology Parameters
Description: Blood samples were collected for the assessment of hematology parameters. The normal ranges for the parameters were: basophil count ([0.00-0.06]*10^9 cells per liter [cells/L]), eosinophil count ([0.02-0.52]*10^9 cells/L), erythrocyte count ([3.8-5.1]*10^12 cells/L), hematocrit (0.35-0.45 proportion of red blood cells in blood), hemoglobin (115-150 g/L), leukocyte count ([3.5-9.5]*10^9 cells/L), lymphocyte count ([1.1-3.2]*10^9 cells/L), monocyte count ([0.1-0.6]*10^9 cells/L), neutrophil count ([1.8-6.3]*10^9 cells/L), platelet count ([125-350]*10^9 cells/L). Number of participants with abnormal hematology parameters are presented.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants | 10 | 15

7. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters
Description: Urine samples were analyzed for glucose, ketones, occult blood and protein by dipstick method. The dipstick test results are read as Negative, Trace, 1+, 2+, 3+, 4+ indicating proportional concentrations in the urine sample. Normal range for dipstick test results are 'negative' results. Urine potential of hydrogen (pH) and specific gravity were also analyzed. pH is measured on a numeric scale of 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Urine specific gravity is a measure of the concentration of solutes in the urine and indicated as ratio of urine density to water density. The normal ranges for pH: 4.8 to 7.4; and for specific gravity: 1.003 to 1.03. Number of participants with abnormal results in any urinalysis parameters are presented.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants | 4 | 11

8. Secondary Outcome: Number of Participants With Injection Site Reaction
Description: Local tolerability as measured by injection site reaction example: induration, erythema, edema, rash, pruritis or pain. Number of participants with any injection site reaction are presented.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants | 0 | 19

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician. Number of participants who had SAEs and non-SAEs are presented.
Time Frame: Up to Day 71
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
Number analyzed (Participants) | 12 | 24
Participants
  SAEs | 0 | 0
  Non-SAEs | 11 | 24

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events were collected from the start of study treatment (Day 1) up to Day 71
Description: SAEs and non-serious adverse events were reported for the Safety Population which comprised of all randomized participants who received at least one dose of study treatment.
Arm/Group | Belimumab 200 mg IV | Belimumab 200 mg SC
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/24
Other Adverse Events (participants affected / at risk) | 11/12 | 24/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 200 mg IV (N=12) | Belimumab 200 mg SC (N=24)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2
Lip blister (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 2
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Injection site hypoaesthesia (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 19
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Vaginal infection (Infections and infestations) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Bacterial test positive (Investigations) | 2 | 4
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood immunoglobulin M decreased (Investigations) | 1 | 3
Blood triglycerides increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 2 | 3
Electrocardiogram T wave abnormal (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 2
Heart rate increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 4
Neutrophil count increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 0 | 4
Urine ketone body present (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 2 | 0
White blood cells urine positive (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Abortion induced (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04136145/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04136145/SAP_001.pdf